CLINICAL TRIAL: NCT00549107
Title: Phase 2 Prospective, Randomized, Double-Blind Pilot Study on Cardiac Output Following Corrective Open Heart Surgery in Children Less Than One Year: Use of Levosimendan Versus Milrinone.
Brief Title: Prophylactic Use of Levosimendan Versus Milrinone in Open Heart Surgery in Infants
Acronym: Levomil
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig Boltzmann Gesellschaft (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-365
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Low Cardiac Output Syndrome
Keywords: low cardiac output syndrome; open heart surgery; infants; Low cardiac output syndrome in infants undergoing corrective open heart surgery
MeSH Terms: conditions — Cardiac Output, Low | interventions — Simendan; Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Levosimendan
- 2 (Active Comparator)
  Interventions: Drug: Milrinone

INTERVENTIONS:
Drug: Levosimendan
  Arms: 1
Drug: Milrinone
  Arms: 2

SUMMARY:
Pediatric patients, especially infants undergoing open heart surgery have a predictable fall in cardiac index 6 to 18 hours after surgery, the so-called low cardiac output syndrome (LCOS). Patients, who have LCOS require more monitoring, more medication and a longer stay in intensive care unit. To prevent LCOS the phosphodiesterase inhibitor milrinone is routinely used during the first 24 hours after surgery. Levosimendan, a calcium- sensitizer improves cardiac muscle contractile force, vascular smooth muscle relaxation and coronary blood flow through calcium sensitization of the myocardial contractile filaments and opening of potassium channels without increasing oxygen consumption of the heart muscle cells. As the myocardium of infants is more calcium dependent than in later life, levosimendan should be of special benefit in this age group. The purpose of this study is to investigate whether levosimendan is superior to milrinone in preventing LCOS in infants after corrective open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age younger than one year
* corrective open heart surgery with biventricular repair, except tetralogy of fallot

Exclusion Criteria:

* Missing written consent of parents
* Weight less than 3 kg
* preoperative LCOS
* gestational age less than 36 weeks
* preexisting renal failure
* preexisting thrombopenia
* preoperative cardiopulmonary resuscitation
* preoperative use of milrinone or levosimendan

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2007-09

PRIMARY OUTCOMES:
Cardiac output measured by a transesophageal probe | 48 hours

SECONDARY OUTCOMES:
Changes in mixed venous saturation | 48 hours
Serum lactate levels | 48 hours
Cardiac output and ventricular function assessed by echocardiography | 48 hours
Mean arterial, left atrial and central venous pressure | 48 hours
Need of catecholamines assessed with the inotropic score | 48 hours
Urine output | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Lechner, MD, Principal Investigator — Children´s Heart Center Linz; Hans Gombotz, MD, PHD, Study Director — General Hospital Linz, Ludwig Boltzmann Gesellschaft; Anna Hofer, MD, Principal Investigator — General Hospital Linz; Gerald Tulzer, MD, PHD, Study Chair — Children´s Heart Center Linz
Locations (1):
- Children´s Heart Center Linz, Linz, Austria

REFERENCES:
- [Background] Wernovsky G, Wypij D, Jonas RA, Mayer JE Jr, Hanley FL, Hickey PR, Walsh AZ, Chang AC, Castaneda AR, Newburger JW, Wessel DL. Postoperative course and hemodynamic profile after the arterial switch operation in neonates and infants. A comparison of low-flow cardiopulmonary bypass and circulatory arrest. Circulation. 1995 Oct 15;92(8):2226-35. doi: 10.1161/01.cir.92.8.2226. PMID 7554206
- [Background] Hoffman TM, Wernovsky G, Atz AM, Kulik TJ, Nelson DP, Chang AC, Bailey JM, Akbary A, Kocsis JF, Kaczmarek R, Spray TL, Wessel DL. Efficacy and safety of milrinone in preventing low cardiac output syndrome in infants and children after corrective surgery for congenital heart disease. Circulation. 2003 Feb 25;107(7):996-1002. doi: 10.1161/01.cir.0000051365.81920.28. PMID 12600913
- [Background] Turanlahti M, Boldt T, Palkama T, Antila S, Lehtonen L, Pesonen E. Pharmacokinetics of levosimendan in pediatric patients evaluated for cardiac surgery. Pediatr Crit Care Med. 2004 Sep;5(5):457-62. doi: 10.1097/01.pcc.0000137355.01277.9c. PMID 15329162
- [Background] Egan JR, Clarke AJ, Williams S, Cole AD, Ayer J, Jacobe S, Chard RB, Winlaw DS. Levosimendan for low cardiac output: a pediatric experience. J Intensive Care Med. 2006 May-Jun;21(3):183-7. doi: 10.1177/0885066606287039. PMID 16672640
- [Background] Namachivayam P, Crossland DS, Butt WW, Shekerdemian LS. Early experience with Levosimendan in children with ventricular dysfunction. Pediatr Crit Care Med. 2006 Sep;7(5):445-8. doi: 10.1097/01.PCC.0000235251.14491.75. PMID 16885788